CLINICAL TRIAL: NCT00001159
Title: Natural History of Thyroid Function Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 770002; 77-DK-0002
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01-09

CONDITIONS: Hyperthyroidism; Hypothyroidism; Grave's Disease
Keywords: Hyperthyroidism; Hypothyroidism; Grave's Disease; Natural History; Thyroid-Stimulating Hormone Secreting Pituitary Ad
MeSH Terms: conditions — Hyperthyroidism; Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid disorders: Patients with thyroid disorders

SUMMARY:
Participants in this study will be patients diagnosed with or suspected to have a thyroid function disorder. These conditions may include: hypothyroidism, hyperthyroidism, thyroid hormone resistance, Graves' Dermopathy, and thyroid-stimulating hormone (TSH) secreting pituitary adenomas.

The main purpose of this study is to further understand the natural history, clinical presentation, and genetics of thyroid function disorders. Many of the tests performed are in the context of standard medical care that is offered to all patients with thyroid function disorders. In addition, blood and tissue samples may be taken for research and genetic studies....

DETAILED DESCRIPTION:
Patients with thyroid function abnormalities (hyperthyroidism, hypothyroidism) are studied and treated in this protocol. Patients undergo routine history and physical examination, standard endocrine blood and urine tests, a standard TRH test, thyroid nuclear medicine scans, thyroidal radioiodine (RAI) or technetium (99mTc) uptake measurements, as well as X-ray, computed tomography (CT) or magnetic resonance imaging (MRI) studies or other standard diagnostic procedures, as clinically indicated.

The goals of this study are:

* 1. To understand the pathophysiology and various causes of thyroid function abnormalities (e.g., hyperthyroidism, hypothyroidism).
* 2. To longitudinally follow the effects of standard therapies for patients with abnormal thyroid functions.
* 3. To create a repository of clinical data and biospecimens for future research of thyroid disorders.

Our objective will be accomplished by obtaining clinical data and biospecimens during standard care procedures and tests performed on enrolled subjects being evaluated as an outpatient in the clinic or as an inpatient at the NIH Clinical Center.

ELIGIBILITY:
* INCLUSION CRITERIA:

The categories of subjects eligible to participate in this study include:

1. Patients with known or suspected thyroid abnormalities (e.g. hypothyroidism, hyperthyroidism, extreme iodine deficiency, and inherited forms of hypothyroidism resulting from abnormalities in the expression of genes coding for the TSH- beta subunit, Pax-8, TTF-2, Pit-I, Tg, PDS, and NIS.
2. Patients with thyroid function test (TFT) abnormalities due to:

   * Non-thyroidal illness
   * Abnormalities of serum TH binding proteins leading to euthyroid hyperthyroxinemia or hypotriiodothyronemia.
   * Genetic deficiency of thyroxine-binding globulin (TBG).
   * Antibodies to mouse immunoglobulins leading to an artifactual elevation in the TSH ultrasensitive ("3rd generation") assay which may mimic "inappropriate" secretion of TSH.

Inclusion and exclusion criteria for each group of subjects are given below.

Patients with known or suspected thyroid abnormalities will be eligible to p rticipate if the individual meets all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Male or female, aged 6 months+.

Hyperthyroid states include but are not restricted to:

1. Graves' disease (GD) thought to result from thyroid-stimulating immunoglobulins (TSIg's), a subclass of which also stimulate eye muscle and fatty tissue producing exophthalmos (Graves' ophthalmopathy), as well as the skin in the pretibial area causing pretibial myxedema (Graves' dermopathy);
2. Subacute thyroiditis (SAT), a painful inflammation thought to result from viral infection with Coxsackie, as well as other viruses;
3. Silent thyroiditis, a painless inflammation thought to result from autoimmune attack of thyrocytes by antimicrosomal antibodies directed against thyroid peroxidase (TPO), as well as antithyroglobulin(anti-Tg) antibodies;
4. Single or multiple hyperfunctioning thyroid nodules of unknown etiology, probably resulting from the activation of certain thyroid oncogenes and/or growth factors, such as the thyrotropin (TSH) receptor (TSHR) and the a-subunit of the G protein (Ga);
5. Iodide-induced hyperthyroidism of unknown etiology;
6. Surreptitious administration of thyroid hormone (TH), usually present in patients with underlying psychiatric disease or occasionally related to patients with obesity and other eating disorders
7. Trophoblastic neoplasms, thought to result from high levels of hCG secretion, which, because of its structural similarity to TSH, causes "spillover" of action at the TSHR level;
8. "Inappropriate" secretion of TSH, which may be present either in patients with TSH- producing pituitary tumors (TSHomas) or from a non-neoplastic cause, i.e. pituitary resistance to the action of thyroid hormone (3,4).

Hypothyroid states include but are not restricted to:

1. Primary (or thyroidal) hypothyroidism, usually resulting from auto-antibodies to thyroid proteins, such as antimicrosomal antibodies to TPO usually associated with lymphocytic (Hashimoto's) thyroiditis (HT) or atrophic thyroiditis, or blocking antibodies to the TSHR, usually in the context of non-goitrous hypothyroidism;
2. Secondary (or pituitary) hypothyroidism, usually resulting from tumors of the pituitary of non-thyrotropic origin such, as growth hormone (GH)-secreting tumors or prolactinomas;
3. Tertiary (or hypothalamic) hypothyroidism, usually resulting from a deficiency in the hypothalamic hormone thyrotropin-releasing hormone (TRH), either of unknown etiology or secondary to a pituitary tumor;
4. Bio-inactive TSH, either relating to an endogenous abnormality of hypothalamic hormones or secondary to pituitary tumors (and usually related to abnormal glycosylation patterns of the TSH molecule);
5. Generalized resistance to thyroid hormone (RTH), a disease which has been shown to be due to abnormalities in the TH receptor, c-erbA-beta (or TR- beta).

The above are the principal disorders under study, but we may also investigate other abnormalities, such as extreme iodine deficiency, and inherited forms of hypothyroidism resulting from abnormalities in the expression of genes coding for the TSH- beta subunit, Pax-8, TTF-2, Pit-I, Tg, PDS, and NIS (among others).

EXCLUSION CRITERIA:

There are no exclusion criteria for subjects with known or suspected thyroid abnormalities.

Ages: 6 Months to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: anyone meeting eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 1977-02-01 (Actual)

PRIMARY OUTCOMES:
evaluation of thyroid disorders | ongoing
  Patients undergo routine history and physical examination, standard endocrine blood and urine tests, a standard TRH test, thyroid nuclear medicine scans, thyroidal radioiodine (RAI) or technetium (99mTc) uptake measurements, as well as X-ray, computed tomography (CT) or magnetic resonance imaging (MRI) studies or other standard diagnostic procedures, as clinically indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Sriram M Gubbi, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Subject level data will be shared upon request after appropriate collaboration agreements are in place.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1977-DK-0002.html